CLINICAL TRIAL: NCT00722124
Title: S-Adenosyl-L-Methionine (SAMe) for Smoking Abstinence
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Pharmavite LLC (Industry)
Responsible Party: Amit Sood, M.D., Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 07-006365; 07-006604
Record Dates: First submitted 2008-07-23; First posted 2008-07-25 (Estimated); Results first posted 2011-09-09 (Estimated); Last update posted 2011-09-09 (Estimated); Status verified 2011-08

CONDITIONS: Tobacco Dependence
Keywords: tobacco use; cigarettes; smokers
MeSH Terms: conditions — Tobacco Use Disorder; Tobacco Use | interventions — S-Adenosylmethionine; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- SAMe 800 (Active Comparator): Each subject randomized to this arm will take a 400 mg pill of SAMe and one matching placebo pill in the AM and again in the PM
  Interventions: Drug: S-Adenosyl-L-Methionine
- SAMe 1600 (Active Comparator): Each person randomized to this arm will take 2 400 mg pills of SAMe in the AM and again in the PM
  Interventions: Drug: S-Adenosyl-L-Methionine
- Placebo (Placebo Comparator): Each subject randomized to this arm will take 2 placebo pills in the AM and again in the PM
  Interventions: Other: placebo

INTERVENTIONS:
Drug: S-Adenosyl-L-Methionine — 800 mg dose per day for 8 weeks
  Other Names: SAMe
  Arms: SAMe 800
Drug: S-Adenosyl-L-Methionine — 1600 mg per day for 8 weeks
  Other Names: SAMe
  Arms: SAMe 1600
Other: placebo — 4 pills (2 in the AM and 2 in the PM) of placebos for 8 weeks
  Other Names: sugar pill
  Arms: Placebo

SUMMARY:
Cigarette smoking is of great public health importance and is the single most important preventable cause of morbidity, mortality and excess health care costs in the United States. After a steady decline for the last 50 years, the prevalence of tobacco use in the United States has reached a plateau of approximately 21%. Currently available treatments among adults are not efficacious for all tobacco users. New pharmacologic agents thus need to be continually developed and tested.

The release of dopamine in the nucleus accumbens is one of the key components of the pleasurable and rewarding effects of nicotine. Drugs that increase monoamine neurotransmitter availability (particularly dopamine and norepinephrine) are likely to increase the reward function and thus ameliorate withdrawal symptoms. S-Adenosyl-L-Methionine (SAMe), the primary methyl donor for the central nervous system (CNS), donates methyl groups towards presynaptic synthesis of CNS monoamine neurotransmitters. By facilitating the synthesis of dopamine and norepinephrine in the brain, SAMe is likely to ameliorate the symptoms of nicotine withdrawal, thus improving tobacco abstinence rates in smokers who are trying to stop smoking. SAMe is well tolerated and is available over-the-counter.

To date, no prospective clinical trial evaluating the efficacy of SAMe for the treatment of tobacco dependence has been published. We propose to evaluate the efficacy of SAMe for increasing smoking abstinence and decreasing nicotine withdrawal symptoms in a randomized, blinded, placebo-controlled, three-arm, parallel-group, dose-ranging phase II clinical trial. Participants (N=120) will be randomly assigned to one of the three groups, and will receive an 8-week course of SAMe 800-mg per day, 1600-mg per day, or a matching placebo. This study is anticipated to provide the data needed to develop a larger randomized controlled clinical trial submitted through the R01 funding mechanism, if the results appear promising.

DETAILED DESCRIPTION:
In this study, after consenting, subject is screened for study eligibility. If they pass the study screen, they are randomized to study drug (800 mg/day of SAMe, 1600 mg/day of SAMe or placebo-look-alike). Subjects will stay on their assigned dose for 8 weeks with weekly (visits 3-6) or biweekly (visits 7-8) clinic visits. After the 8 weeks of medication, they will receive a phone visit at week 16 and then a final visit at week 24. Study participation ends at the week 24 visit. During study participation, subjects will undergo counseling at every study visit based on the counseling manual, Smoke Free and Living It. They will also keep diaries (record of daily withdraw symptoms and tobacco use) for the 8 weeks while on study medication. At each study visit, smoking and safety outcomes are measured.

ELIGIBILITY:
Inclusion Criteria:

* Is at least 18 years of age;
* Has smoked more than 10 cigarettes/day for ≥6 months;
* Is willing to make a quit attempt;
* Is able to participate fully in all aspects of the study;
* Has been provided with, understand, and have signed the informed consent.
* Is in good health as determined by the physician investigator.

Exclusion Criteria:

* Is clinically significant levels of current depression as assessed by CESD (Score >16) and determined by the physician; or have a life-time diagnosis of bipolar disorder, schizophrenia or dementia as determined by physician investigator;
* Has an unstable medical condition.
* Is using other tobacco product and the primary use is NOT cigarettes.
* Is currently (within the past 30-days) using antipsychotics or antidepressants;
* Is currently (within the past 30-days) using any treatments for tobacco dependence (i.e., behavioral therapy, nicotine replacement therapy, bupropion SR, clonidine, or nortriptyline);
* Is currently using another investigational drug at the time of study enrollment;
* Is currently (within the past 30 days) using an herbal product or dietary supplement for tobacco abstinence;
* Has recent history (in the past 3-months) of alcohol abuse or dependence as assessed by the CAGE questionnaire and study investigators;
* Has a recent history of drug abuse as assessed by physician interview;
* Is pregnant, lactating, or of child bearing potential, likely to become pregnant during the medication phase and not willing to use a reliable form of contraception. Reliable forms of contraception include diaphragm or condom (with spermicidal), injections, intrauterine device [IUD], surgical sterilization and abstinence;
* Is a history of any major cardiovascular events in the past 3-months including unstable angina, acute MI or coronary angioplasty;
* Has clinically significant acute or chronic progressive or unstable neurologic, hepatic, renal, cardiovascular, respiratory or metabolic disease;
* Is currently on medications interacting with SAMe, including but not limited to, antidepressants, MAO inhibitors, levodopa, meperidine, dextromethorphan, pentazocine and tramadol;
* Has another household member or relative participating in the study;
* Has known allergy to SAMe.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2008-09; Primary Completion 2009-12 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amit Sood, M.D., Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic, Rochester, Minnesota
  - Franciscan Skemp HealthCare, La Crosse, Wisconsin

REFERENCES:
- [Derived] Hajizadeh A, Howes S, Theodoulou A, Klemperer E, Hartmann-Boyce J, Livingstone-Banks J, Lindson N. Antidepressants for smoking cessation. Cochrane Database Syst Rev. 2023 May 24;5(5):CD000031. doi: 10.1002/14651858.CD000031.pub6. PMID 37230961

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began on 10/07/08 and completed on 10/01/09. Interested subjects who passed a phone pre-screen were seen at a medical clinic (Mayo Clinic in Rochester, MN and Franciscan Skemp Medical Center in Lacrosse, WI) for consenting and additional study procedures to determine eligibility.
Period: Overall Study
Arm/Group | SAMe 800 | SAMe 1600 | Placebo
Started | 40 | 40 | 40
Completed | 23 | 26 | 20
Not Completed | 17 | 14 | 20

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SAMe 800 | SAMe 1600 | Placebo | Total
Number analyzed (Participants) | 40 | 40 | 40 | 120
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 34 | 40 | 38 | 112
  >=65 years | 6 | 0 | 2 | 8
Age Continuous [Mean (Standard Deviation); unit: years] | 42.1 (16.0) | 40.8 (12.3) | 37.0 (13.6) | 39.9 (14.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 20 | 20 | 57
  Male | 23 | 20 | 20 | 63
baseline smoking rate [Mean (Standard Deviation); unit: cigarettes per day] — Average cigarettes per day at study entry
  cigarettes per day | 19.5 (9.3) | 19.9 (8.4) | 19.5 (8.0) | 19.6 (8.5)

OUTCOME MEASURES:

1. Primary Outcome: 7-day Point Prevalence Smoking Abstinence at End of Treatment (Week 8)
Description: 7-day point prevalence smoking abstinence biochemically confirmed (expired carbon monoxide <8ppm)
Time Frame: 8 weeks
Population: Analysis was performed using intention to treat(ITT). Subjects who discontinued study participation were assumed to be smoking.
Measure: Number; unit: participants
Arm/Group | SAMe 800 | SAMe 1600 | Placebo
Number analyzed (Participants) | 40 | 40 | 40
participants | 7 | 5 | 7
Statistical Analysis 1: Comparison: SAMe 800 vs Placebo; Data were compared between treatment groups using Fisher's Exact test; Test type: Superiority or Other; p = 0.615, Fisher Exact; 1 sided
Statistical Analysis 2: Comparison: SAMe 1600 vs Placebo; Data were compared between treatment groups using Fisher's Exact test; Test type: Superiority or Other; p = 0.826, Fisher Exact; 1 sided

ADVERSE EVENTS:
Arm/Group | SAMe 800 | SAMe 1600 | Placebo
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 7/40 | 12/40 | 6/40
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SAMe 800 (N=40) | SAMe 1600 (N=40) | Placebo (N=40)
abdominal pain (Gastrointestinal disorders) | 2 | 5 | 1
nausea (Gastrointestinal disorders) | 2 | 2 | 2
headache (General disorders) | 2 | 0 | 2
diarrhea (Gastrointestinal disorders) | 0 | 3 | 0
insomnia (General disorders) | 0 | 1 | 1
anorexia (Metabolism and nutrition disorders) | 0 | 1 | 0
confusion (General disorders) | 0 | 1 | 0
constipation (Gastrointestinal disorders) | 1 | 0 | 0
dizziness (General disorders) | 0 | 0 | 1
drowsiness/fatigue (General disorders) | 1 | 0 | 0
flatulence (Gastrointestinal disorders) | 0 | 1 | 0
heartburn (Gastrointestinal disorders) | 0 | 1 | 0
vivid dreams (General disorders) | 0 | 0 | 1
vomiting (Gastrointestinal disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No